CLINICAL TRIAL: NCT01278290
Title: Triptorelin Acetate Utilization for the Early Diagnosis of Central Precocious Puberty (CPP) in Girls.
Brief Title: Comparative Validation of the Triptorelin Test for the Diagnosis of CPP in Girls
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Niños R. Gutierrez de Buenos Aires (Other)
Responsible Party: Principal Investigator, Analía Freire, Pediatric Endocrinology, PhD, Hospital de Niños R. Gutierrez de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HNinosBuenosAires-Triptorelin
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Central Precocious Puberty; Sexual Precocity
Keywords: Triptorelin acetate; precocious puberty; premature thelarche; GnRH analog; Diagnostic validation study
MeSH Terms: conditions — Puberty, Precocious

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triptorelin test AND LHRH test (Active Comparator): Patients undergo two tests with a test interval of at least 15 days
  Interventions: Diagnostic Test: Triptorelin acetate and Gonadorelin acetate
- LHRH test AND Triptorelin test (Active Comparator): Patients undergo two test with a test interval of al least 15 days.
  Interventions: Diagnostic Test: Gonadorelin acetate and Triptorelin acetate

INTERVENTIONS:
Diagnostic Test: Triptorelin acetate and Gonadorelin acetate — Triptorelin acetate test, using aqueous 0.1 mg/m2 subcutaneous. Gonadorelin test using 100 ug intravenous.
  Arms: Triptorelin test AND LHRH test
Diagnostic Test: Gonadorelin acetate and Triptorelin acetate — Gonadorelin acetate intravenous 100 ug. Triptorelin acetate 100 ug/m2.
  Arms: LHRH test AND Triptorelin test

SUMMARY:
The aim of the study is to determine the specificity, sensitivity and diagnostic efficiency of the Triptorelin Test in the assessment of CPP compared to GnRH test as gold standard.

Hypothesis: Aqueous Triptorelin Acetate is so efficient as GnRH to CPP assessment.

Study population are girls with suspicious clinical features of precocious puberty

DETAILED DESCRIPTION:
GnRH stimulation is the gold standard to distinguish between isolated premature thelarche (PT) and CPP. However, intravenous GnRH for testing is not fully available in all countries. To evaluate the diagnostic accuracy of a novel Triptorelin-test in the assessment of CPP compared to the GnRH test, a validation study was performed. Girls who presented thelarche with accelerated growth and/or advanced bone age were included. All girls underwent the two tests in a randomized order. CPP was ascertained according to LH response under GnRH (gold standard test).

ELIGIBILITY:
Inclusion Criteria:

* premature thelarche and/or
* accelerated growth velocity (above 90 percentile)
* advanced bone age at least 1.5 year in relation to chronological age.

Exclusion Criteria:

* contact with sources of exogenous estrogens in the last four months previous to evaluation,
* suspicion of peripheral precocious puberty,
* previous central nervous system illness or suspicion of organic central precocious puberty.

Ages: 3 Years to 8 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2009-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
LH | 3 hs
  Levels of LH are measured at T 0 (before) and T 3 h y T 24 h (after) Triptorelin stimulation.
Estradiol | 24 hs
  Levels of Estradiol are measured at T 0 (before) and T 3 h y T 24 h (after) Triptorelin stimulation.

SECONDARY OUTCOMES:
FSH | 3 hs
  Levels of FSH are measured at T 0 (before) and T 3 h y T 24 h (after) Triptorelin stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Maria G Ropelato, PhD, Study Director — División de Endocrinología, Hospital de Niños Ricardo Gutierrez, Buenos Aires, Argentina; Analía V Freire, MD, Principal Investigator — División de Endocrinología, Hospital de Niños Ricardo Gutiérrez, Buenos Aires, Argentina
Locations (1):
- Hospital de Niños Ricardo Gutierrez, División de Endocrinología, Buenos Aires, Argentina